CLINICAL TRIAL: NCT06625658
Title: Evaluation of Direct 3D Printed Clear Aligners for Treatment of Maxillary Anterior Crowding:(Clinical Trial)
Brief Title: Evaluation of DPA for Treatment of Upper Anterior Crowding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samia Omar (Other Government)
Responsible Party: Sponsor-Investigator, Samia Omar, dentist, Faculty of Dental Medicine for Girls
Organization: Faculty of Dental Medicine for Girls (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-109-2- N
Record Dates: First submitted 2024-09-29; First posted 2024-10-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Correction of Upper Crowding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- clear aligner therapy (Experimental)
  Interventions: Device: Direct printed clear aligners

INTERVENTIONS:
Device: Direct printed clear aligners — chang aligner every 10 days

SUMMARY:
Evaluation of effectiveness of direct printed clear aligner in relive crowding in maxillary incisor

DETAILED DESCRIPTION:
The present study will be performed to evaluate the effectiveness of direct 3D-printed aligners in the treatment of maxillary anterior teeth crowding

ELIGIBILITY:
Inclusion Criteria:

* Adult paients .age 18-25y. patients with mild to moderate upper anterior crowding (1mm_6mm)
* Healthy compliant and motivated patient. full dentition except wisdom teeth.

Exclusion Criteria:

* Previous orthodontic treatments. Any systemic disease, pregnancy, or lactating females, with a pocket depth of more than 5mm.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correction of Maxillary Anterior Teeth Crowding according to little irregularity index | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sara M .Hosny El kabbany, assistant professor, Principal Investigator — Study Principal Investigator Al azhar universty
Locations (1):
- Al Azhar University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No